CLINICAL TRIAL: NCT04354545
Title: Treatment of Ocular Discomfort in Glaucoma Patients Using Multiple Topical Medications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Benjamin B. Bert, MD, Health Sciences Assistant Professor, University of California, Los Angeles
Other Study IDs: 19-000843
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma; Ocular Surface Disease
Keywords: glaucoma; xiidra™; ocular surface discomfort
MeSH Terms: conditions — Glaucoma | interventions — lifitegrast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Xiidra (Lifitegrast ophthalmic solution) 5% applied to both eye (OU) for 12 weeks
  Interventions: Drug: Xiidra (Lifitegrast ophthalmic solution) 5%

INTERVENTIONS:
Drug: Xiidra (Lifitegrast ophthalmic solution) 5% — FDA approved lifitegrast opthalmic solution eye drop
  Other Names: Lifitegrast ophthalmic solution; SAR-1118

SUMMARY:
To evaluate glaucoma patients' response to treatment with Xiidra, an FDA-approved drug for ocular surface discomfort, which will be prescribed as standard of care treatment.

DETAILED DESCRIPTION:
To assess glaucoma patients' response to treatment with Xiidra (Lifitegrast ophthalmic solution) 5% for ocular surface discomfort caused, in part, by topical glaucoma antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Currently using one or more topical glaucoma antihypertensives
* Self-described symptoms of ocular surface discomfort
* Xiidra is being prescribed as part of the subject's standard care

Exclusion Criteria:

* History of glaucoma filtration surgery, history of ocular surface surgery (pterygium, conjunctivoplasty, etc.),
* current use of topical cyclosporine
* current use of topical steroids
* incisional ocular surgery within 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Glaucoma patients suffering from ocular surface discomfort
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 12 in corneal fluorescein staining score | From baseline to Week 12
  Change in corneal fluorescein staining score
Change from baseline to week 12 in eye dryness score (EDS) | From baseline to Week 12
  Change in eye dryness score (EDS)
Change from baseline to week 12 in ocular surface disease index (OSDI) questionnaire score | From baseline to Week 12
  Change in ocular surface disease index (OSDI) questionnaire score

SECONDARY OUTCOMES:
Change at intermediate week visits in corneal fluorescein staining score | From baseline and at weeks 2, 6, and 12
  Change in corneal fluorescein staining score
Change at intermediate week visits in eye dryness score (EDS) | From baseline and at weeks 2, 6, and 12
  Change in eye dryness score (EDS)
Change at intermediate week visits in ocular surface disease index (OSDI) questionnaire score | From baseline and at weeks 2, 6, and 12
  Change in ocular surface disease index (OSDI) questionnaire score
Changes in the subcategories of ocular surface disease index (OSDI) questionnaire score at intermediate week visits | From baseline and at weeks 2, 6, and 12
  Change in subcategory scores of ocular surface disease index (OSDI) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Doheny Eye Center UCLA, Fountain Valley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT04354545/ICF_000.pdf